CLINICAL TRIAL: NCT01959672
Title: A Phase II Study of Neoadjuvant Chemotherapy With and Without Immunotherapy to CA125 (Oregovomab) Followed by Hypofractionated Stereotactic Radiotherapy & Concurrent HIV Protease Inhibitor Nelfinavir in Locally Advanced Pancreatic Cancer
Brief Title: Chemotherapy, Stereotactic Body Radiation Therapy & Nelfinavir Mesylate in Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0441-13-FB; NCI-2013-02273 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2013-02118 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2012-00835 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Adenocarcinoma; Resectable Pancreatic Carcinoma; Stage I Pancreatic Cancer; Stage IA Pancreatic Cancer; Stage IB Pancreatic Cancer; Stage II Pancreatic Cancer; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer; Stage III Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; dehydroftorafur; Gemcitabine; Leucovorin; Nelfinavir; oregovomab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, oregovomab, SBRT, surgery) (Experimental): CHEMOTHERAPY: Patients receive gemcitabine hydrochloride IV, leucovorin calcium IV over 30 minutes, and fluorouracil IV over 24 hours on days 1 and 8. Treatment repeats every 3 weeks for 7 courses.
  IMMUNOTHERAPY: Patients with CA125 level >= 10 receive oregovomab IV over 15-30 minutes on day 15. Treatment repeats every 3 weeks for 3 courses (weeks 1, 4, 7) and post- radiation therapy for 1 course (week 14). Patients may receive an additional 3 courses concurrently with chemotherapy upon recovery from surgery based on CA125 level. Patients also receive nelfinavir mesylate PO BID for 5 weeks beginning on day 15 of week 9.
  STEREOTACTIC RADIATION THERAPY: Beginning in week 11, patients undergo SBRT in 5 fractions over 5 consecutive days. Upon completion of radiation therapy, patients resume nelfinavir mesylate for 14 days (week 12-13). Patients without metastasis and with resectable disease undergo surgery in week 17-18.
  Interventions: Procedure: 4-Dimensional Computed Tomography; Drug: Fluorouracil; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Nelfinavir Mesylate; Biological: Oregovomab; Radiation: Stereotactic Body Radiation Therapy; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: 4-Dimensional Computed Tomography — Correlative studies
  Other Names: 4D Computed Tomography; 4DCT; Time-Resolved CT Data Acquisition
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Nelfinavir Mesylate — Given PO
  Other Names: AG1343; Viracept
Biological: Oregovomab — Given IV
  Other Names: B43.13; MoAb B43.13; Monoclonal Antibody B43.13; OvaRex; OvaRex Monoclonal Antibody B43.13
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SBRT
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection

SUMMARY:
This phase II trial studies how well combination chemotherapy with or without oregovomab followed by stereotactic body radiation therapy (SBRT) and nelfinavir mesylate works in treating patients with pancreatic cancer that has spread to nearby organs or tissues. Drugs used in chemotherapy, such as gemcitabine hydrochloride, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as oregovomab, can block tumor growth in different ways by targeting certain cells. Stereotactic body radiation therapy is a specialized radiation therapy that sends x-rays directly to the tumor using smaller doses over several days and may cause less damage to normal tissue. Drugs, such as nelfinavir mesylate, may make tumor cells more sensitive to radiation therapy. Giving combination chemotherapy with or without oregovomab followed by SBRT and nelfinavir mesylate may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of neoadjuvant chemotherapy, (gemcitabine [gemcitabine hydrochloride], leucovorin [leucovorin calcium], fluorouracil [5-FU]) with or without oregovomab, followed by hypofractionated stereotactic radiotherapy (SRT) concurrently with nelfinavir (nelfinavir mesylate) in patients with locally advanced pancreatic cancer that is cancer antigen (CA)125 positive (>= 10) or CA125 negative (< 10).

SECONDARY OBJECTIVES:

I. To assess the safety of neoadjuvant chemotherapy, (gemcitabine, leucovorin, 5-FU) with or without oregovomab, followed by SRT concurrently with nelfinavir in patients with locally advanced pancreatic cancer that is CA125 positive (>= 10) or CA125 negative (< 10).

II. To assess the cellular and humoral immune responses to active immunotherapy with oregovomab/monoclonal antibody in patients with pancreas cancer with CA125 level greater than 10 undergoing chemotherapy and radiation treatments.

TERTIARY OBJECTIVES:

I. To evaluate tumor and organ motion with 4-dimensional (4D) computed tomography (CT) and respiratory gating system.

II. To evaluate the effect of tumor/organ motion on the dosimetry, local control and survival.

III. To evaluate inter- and intra-fractional target motion with Calypso system.

OUTLINE:

CHEMOTHERAPY: Patients receive gemcitabine hydrochloride intravenously (IV), leucovorin calcium IV over 30 minutes, and fluorouracil IV over 24 hours on days 1 and 8. Treatment repeats every 3 weeks for 7 courses.

IMMUNOTHERAPY: Patients with CA125 level >= 10 receive oregovomab IV over 15-30 minutes on day 15. Treatment repeats every 3 weeks for 3 courses (weeks 1, 4, 7) and post- radiation therapy for 1 course (week 14). Patients may receive an additional 3 courses concurrently with chemotherapy upon recovery from surgery based on CA125 level. Patients also receive nelfinavir mesylate orally (PO) twice daily (BID) for 5 weeks beginning on day 15 of week 9.

STEREOTACTIC RADIATION THERAPY: Beginning in week 11, patients undergo SBRT in 5 fractions over 5 consecutive days. Upon completion of radiation therapy, patients resume nelfinavir mesylate for 14 days (week 12-13). Patients without metastasis and with resectable disease undergo surgery in week 17-18.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the pancreas; patients have resectable borderline resectable disease, or unresectable disease with no evidence of distant metastases or peritoneal disease; the maximum dimension of the tumor must be =< 10 cm
* Karnofsky performance status of 60% or better
* Patients who received chemotherapy > 5 years ago for malignancies other than pancreatic cancer are eligible, provided that chemotherapy was completed > 5 years ago and that there is no evidence of the second malignancy at the time of study entry
* Patients who received radiation therapy > 5 years ago for malignancies other than pancreatic cancer and whose radiation therapy field is not overlapping with the 20% isodose line of current radiation field are eligible, provided that radiation therapy was completed > 5 years ago and that there is no evidence of the second malignancy at the time of study entry
* All malignant disease must be able to be encompassed within a single irradiation field
* All patients must have radiographically assessable disease
* Absolute neutrophil count (ANC) greater than or equal to 1500/uL
* Platelet count greater than or equal to 100,000/uL
* Serum creatinine less than or equal to 2.0 mg/dL
* Total bilirubin less than or equal to 2.0 mg/dL in the absence of biliary obstruction; if the patient has biliary obstruction, biliary decompression will be required; either endoscopic placement of biliary stent (7 French or greater) or percutaneous transhepatic drainage are acceptable; once biliary drainage has been established, institution of gemcitabine therapy may proceed when the total bilirubin falls to =< 4.0 mg/dL; patients with biliary or gastroduodenal obstruction must have drainage or surgical bypass prior to starting chemoradiation
* The patient must be aware of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts
* No prior therapy with the exception of 1 cycle of chemotherapy based on current diagnosis and clinical condition
* Patients must have CA125 level >= 10 to participate in the immunotherapy aspect of the trial and receive oregovomab; if the patient has CA125 >= 10 who is not eligible to receive oregovomab (e.g. allergic to the drug) but is eligible for the rest of treatment, this patient should be accrued to the part of protocol without oregovomab

Exclusion Criteria:

* Patients who cannot undergo staging laparoscopy; for example, this may include patients with a prior history of multiple abdominal operations in which laparoscopy may not be technically feasible or potentially harmful; the patient is eligible if they have a common bile duct stent adjacent to the tumor that may be used as an internal marker, or if the patient has already had a staging laparoscopy without marker implantation and the markers can be implanted (by interventional radiology) prior to the beginning of radiation therapy
* Patients with a known allergy to murine proteins or have had a documented anaphylactic reaction or allergy to any of chemotherapy agents used in this protocol, oregovomab, or to antiemetics appropriate for administration in conjunction with protocol-directed therapy
* Uncontrolled inter-current illness including, but not limited to ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure, unstable angina pectoris, or serious, uncontrolled cardiac arrhythmia, that might jeopardize the ability of the patient to receive the therapy program outlined in this protocol with reasonable safety
* Pregnant and nursing women are excluded from this study
* Patients with prior malignancy will be excluded except for adequately treated basal cell or squamous cell skin cancer, adequately treated noninvasive carcinomas, or other cancers from which the patient has been disease-free for at least 5 years
* Patients with active duodenal ulcer or bleeding or history of a gastrointestinal fistula or perforation or other significant bowel problems (severe nausea, vomiting, inflammatory bowel disease and significant bowel resection)
* Patients with known human immunodeficiency virus (HIV) infection, or hepatic insufficiency
* Patients who cannot take oral medications
* Patients may not be receiving or have received any other investigational agents during/or within 1 month prior to treatment with oregovomab or nelfinavir
* Patients with an active autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus [SLE], ulcerative colitis, Crohn's disease, multiple sclerosis [MS], ankylosing spondylitis)
* Patients with a recognized acquired, hereditary, or congenital immunodeficiency disease including cellular immunodeficiency's, hypogammaglobulinemia or dysgammaglobulinemia
* Patients receiving the following drugs that are contraindicated with nelfinavir (NFV) (VIRACEPT) will be excluded if they cannot be change or discontinued; drugs that should not be coadministered with Viracept:

  * Antiarrhythmics: amiodarone, quinidine
  * Antimycobacterial: rifampin
  * Ergot derivatives: dihydroergotamine, ergonovine, ergotamine, methylergonovine
  * Herbal products: St. John's wort (hypericum perforatum)
  * 3-hydroxy-3-methyl-glutaryl (HMG)-acetyl coenzyme A (CoA) reductase inhibitors: lovastatin, simvastatin
  * Neuroleptic: pimozide
  * Sedative/hypnotics: midazolam, triazolam
* Patients receiving the following drugs will be clinically evaluated as to whether dosage/medication can be changed to permit patient on study:

  * Anti-convulsants: carbamazepine, phenobarbital
  * Anti-convulsant: phenytoin; phenytoin plasma/serum concentrations should be monitored; phenytoin dose may require adjustment to compensate for altered phenytoin concentration
  * Anti-mycobacterial: rifabutin; it is recommended that the dose of rifabutin be reduced to one-half the usual dose when administered with VIRACEPT; 1250 mg BID is the preferred dose of VIRACEPT when coadministered with rifabutin
  * Erectile dysfunction agent: sildenafil; sildenafil shall not exceed a maximum single dose of 25 mg in a 48 hour period
  * HMG-CoA reductase inhibitor: atorvastatin; use lowest possible dose of atorvastatin with careful monitoring, or consider other HMG-CoA reductase inhibitors such as pravastatin or fluvastatin in combination with VIRACEPT
  * Immunosuppressants: cyclosporine, tacrolimus, sirolimus
  * Narcotic analgesic: methadone; dosage of methadone may need to be increased when coadministered with VIRACEPT
  * Oral contraceptive: ethinyl estradiol; alternative or additional contraceptive measures should be used when oral contraceptives and VIRACEPT are coadministered
  * Macrolide antibiotic: azithromycin; dose adjustment of azithromycin is not recommended, but close monitoring for known side effects such as liver enzyme abnormalities and hearing impairment is warranted

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-09-06 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi Lin, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Oregovomab, SBRT, Surgery)
Started | 11
Completed | 10
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, Oregovomab, SBRT, Surgery)
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 65 [45 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progressive Disease,
Description: Rate of progressive disease defined as at least a 25% increase in the longest diameter of a lesion, taking as reference the longest diameter recorded since the treatment started. An exact one-sided 90% confidence interval will be constructed round the progressive disease rate.
Time Frame: Up to 4 months
Population: Analysis of the primary endpoint (progression at 4 months) demonstrated that of the ten patients who remained alive, two (20%) had progressed at 4 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Oregovomab, SBRT, Surgery)
Number analyzed (Participants) | 10
Participants | 2

2. Secondary Outcome: Distant Failure-free Survival
Description: Analyzed using Kaplan-Meier plots, medians and ranges.
Time Frame: Date of administration study drug to the date of first appearance of tumor lesions by imaging, or death, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Chemotherapy, Oregovomab, SBRT, Surgery)
Number analyzed (Participants) | 11
months | 11 [7 to 15]

3. Secondary Outcome: Overall Survival
Description: Analyzed using Kaplan-Meier plots, medians and ranges.
Time Frame: Date of first of study drug to the date of death, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Chemotherapy, Oregovomab, SBRT, Surgery)
Number analyzed (Participants) | 11
months | 14.4 [12 to 18]

4. Secondary Outcome: Surgical Complete Resection (Negative Margin) Rate
Description: The percentage of patients who will undergo R0 resection
Time Frame: Up to week 18
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Chemotherapy, Oregovomab, SBRT, Surgery): CHEMOTHERAPY: Patients receive gemcitabine hydrochloride IV, leucovorin calcium IV over 30 minutes, and fluorouracil IV over 24 hours on days 1 and 8. Treatment repeats every 3 weeks for 7 courses.
  IMMUNOTHERAPY: Patients with CA125 level >= 10 receive oregovomab IV over 15-30 minutes on day 15. Treatment repeats every 3 weeks for 3 courses (weeks 1, 4, 7) and post- radiation therapy for 1 course (week 14). Patients may receive an additional 3 courses concurrently with chemotherapy upon recovery from surgery based on CA125 level.
  STEREOTACTIC RADIATION THERAPY: Beginning in week 11, patients undergo SBRT in 5 fractions over 5 consecutive days.
  NELFINAVIR: PO BID for 5 weeks beginning in week 9.
  SURGERY: week 17-18.
Arm/Group | Treatment (Chemotherapy, Oregovomab, SBRT, Surgery)
Number analyzed (Participants) | 10
Participants | 4

5. Secondary Outcome: Tumor Response Rate, Evaluated on the Pathology Specimen
Description: The percentage of patients responding will be summarized using frequencies and percentages. Define poor, intermediate and good response as follows: Score 1-3: poor response to neoadjuvant therapy (still have majority of cancer at the time of surgery) Score 4-6: intermediate response to neoadjuvant therapy (still have moderate amount of cancer at the time of surgery) Score 7-9: good response to neoadjuvant therapy (have minimal amount of residual cancer at the time of surgery)
Time Frame: Up to week 18
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Chemotherapy, Oregovomab, SBRT, Surgery): CHEMOTHERAPY: Patients receive gemcitabine hydrochloride IV, leucovorin calcium IV over 30 minutes, and fluorouracil IV over 24 hours on days 1 and 8. Treatment repeats every 3 weeks for 7 courses.
  IMMUNOTHERAPY: Patients with CA125 level >= 10 receive oregovomab IV over 15-30 minutes on day 15. Treatment repeats every 3 weeks for 3 courses (weeks 1, 4, 7) and post- radiation therapy for 1 course (week 14). Patients may receive an additional 3 courses concurrently with chemotherapy upon recovery from surgery based on CA125 level.
  STEREOTACTIC RADIATION THERAPY: Beginning in week 11, patients undergo SBRT in 5 fractions over 5 consecutive days. Upon completion of radiation therapy, 2-13).
  NELFINAVIR MESYLATE: PO BID for 5 weeks beginning in week 9.
  SURGERY: week 17-18.
Arm/Group | Treatment (Chemotherapy, Oregovomab, SBRT, Surgery)
Number analyzed (Participants) | 4
Participants
  Pathologic poor response | 2
  Pathologic intermediate response | 1
  Pathologic good response | 1

6. Other Pre Specified Outcome: Number of Participants With CA-125-Specific T-cell Signal.
Description: The percentage of patients responding will be summarized using frequencies and percentages.
Time Frame: Baseline to up to week 12
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Chemotherapy, Oregovomab, SBRT, Surgery): CHEMOTHERAPY: Patients receive gemcitabine hydrochloride IV, leucovorin calcium IV over 30 minutes, and fluorouracil IV over 24 hours on days 1 and 8. Treatment repeats every 3 weeks for 7 courses.
  IMMUNOTHERAPY: Patients with CA125 level >= 10 receive oregovomab IV over 15-30 minutes on day 15. Treatment repeats every 3 weeks for 3 courses (weeks 1, 4, 7) and post- radiation therapy for 1 course (week 14). Patients may receive an additional 3 courses concurrently with chemotherapy upon recovery from surgery based on CA125 level.
  STEREOTACTIC RADIATION THERAPY: Beginning in week 11, patients undergo SBRT in 5 fractions over 5 consecutive days.
  NELFINAVIR MESYLATE: PO BID for 5 weeks beginning in week 9.
  SURGERY: week 17-18.
Arm/Group | Treatment (Chemotherapy, Oregovomab, SBRT, Surgery)
Number analyzed (Participants) | 5
Participants | 2

ADVERSE EVENTS:
Time Frame: From the time of informed consent until 30 days after last administration of study medication - approximately 22 weeks
Description: 6 of 9 patients experienced any grade ≥3 adverse event
Arm/Group | Treatment (Chemotherapy, Oregovomab, SBRT, Surgery)
All-Cause Mortality (participants affected / at risk) | 11/11
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Oregovomab, SBRT, Surgery) (N=11)
Anemia (Blood and lymphatic system disorders) | 2 (2) — 2 grade 3
Leukopenia (Investigations) | 6 (6) — 3 grade 3 and 3 grade 4
Thrombocytopenia (Investigations) | 4 (4) — 4 grade 3
Lymphopenia (Investigations) | 4 (4) — 4 grade 3
Reduced ANC (Investigations) | 2 (2) — 2 grade 3 and 4 grade 4
Nausea (Investigations) | 1 (1) — 1 grade 3
Vomiting (Gastrointestinal disorders) | 1 (1) — 1 grade 3
Dehydration (Investigations) | 1 (1) — 1 grade 3
Depression (Investigations) | 1 (1) — 1 grade 3
Somnolence (Renal and urinary disorders) | 1 (1) — 1 grade 3
Hypokalemia (Gastrointestinal disorders) | 1 (1) — 1 grade 3
Hyperkalemia (Infections and infestations) | 1 (1) — 1 grade 3
ALT elevation (Metabolism and nutrition disorders) | 2 (2) — 2 grade 3
AST elevation (Vascular disorders) | 2 (2) — 1 grade 3 and 1 grade 4
Pancreatitis (Investigations) | 1 (1) — 1 grade 3
Pneumonia (Vascular disorders) | 1 (1) — 1 grade 4
Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 grade 4
Urinary tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 grade 3
Sepsis (Metabolism and nutrition disorders) | 1 (1) — 1 grade 4
Pleural effusion (Nervous system disorders) | 1 (1) — 1 grade 4
Sinusitis (Cardiac disorders) | 1 (1) — 1 grade 3
Cardiac disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Oregovomab, SBRT, Surgery) (N=11)
Orthostasis (Investigations) | 1 (1) — 1 grade 1-2
Rash (Investigations) | 1 (1) — 1 grade 1-2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT01959672/Prot_SAP_000.pdf